CLINICAL TRIAL: NCT04961242
Title: Pilot Evaluation of Together for Wellness Website in COVID-19
Acronym: (T4W)
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: California Department of Health Services (Other); University of California, Davis (Other)
Responsible Party: Principal Investigator, Kenneth B. Wells, Professor, University of California, Los Angeles
Other Study IDs: 20-002163
Record Dates: First submitted 2021-07-01; First posted 2021-07-14 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Digital Mental Health Resources (Website) for Coping With Stress and Information
Keywords: digital mental health resources, website, user feedback and evaluation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Together for Wellness digital mental health website — The intervention is a digital mental health resources website that includes multiple, free resources for broad public use. Different categories of resources include information on COVID-19 from CDC, multi-language versions of the UCLA Mindfulness App and other meditation programs, resources for families and social connection, including addressing discrimination or equity, and resource links.

SUMMARY:
This is a pilot evaluation of a set of free digital mental health resources developed for COVID-19 relief in California, with funding for the evaluation by the California Health Care Foundation. The website includes resources to support information on COVID-19, meditation and stress management, resources for parenting resilience, resources for social connection and addressing structural racism, and linkages to resources under the partnering "CalHOPE" website (FEMA funded). The evaluation includes: 1) an invitation from a partnering agency to visit the website and consider the evaluation; 2) a post website visit baseline survey; 3) a follow-up survey 4-6 weeks later; 4) a telephone interview for a subset of participants who agree to the follow-up interview and provide their contact information.

DETAILED DESCRIPTION:
Relevance:

The COVID-19 pandemic has raised awareness of mental health as a primary public health concern. Physical distancing, business and school closures, grief, and stress are aspects of the pandemic with significant mental health consequences. The pandemic has also disproportionately impacted Black, Asian and Pacific Islander, Indigenous, and Latino populations. Concurrent with the pandemic has been a surge in attention on police violence toward Black Americans as well as systemic racism against other groups (Asian) and in other institutions. These stressors are also likely to have substantial mental health consequences. To support addressing these concerns, the state requested development of a website (Together for Wellness) with input from stakeholders across the state, to support dealing with informational needs and stress of diverse stakeholders across the state. In addition, a goal was to obtain user feedback data to understand impact of the website Below are aims for the initial survey, qualitative interview for a subsample, and follow-up survey.

Specific Aims for Initial Survey:

Specific Aim 1: To understand the subjective value of a website of free mental health resources for users of various ethnicities, ages, and who may differ in baseline mental health status and use of mental health services.

Specific Aim 2: To understand the subjective value of a website of free mental health resources for users with various degrees of COVID-related stress.

Specific Aims for Qualitative Interviews:

The broad goal is to use qualitative interviews to more deeply understand the experiences of participants in reviewing the website, their needs for support for themselves, family or community, and ideas for further development of the website. The qualitative interview data will also be linked to their survey data and google analytics data, and de-identified.

Specific Aim 3: To understand the experiences of users who reviewed the website of free mental health resources, using a semi-structured interview guide to examine responses to the website, their needs for support for themselves, family or community, and ideas for improving the website.

Specific Aim 4: To understand how subjective experiences may vary across website users, and to gain insight from participants from various strata (e.g., various race/ethnicity groups, those who live in urban and rural locations, those with various levels of COVID-related stress, and people of different age groups and different gender identities, or other demographics). With stakeholder input, we will select priorities for stratification of sampling (and may increase the number of interviews conducted based on resources available to partnering stakeholder groups through existing contracts that some agencies have with the Mental Health Services Oversight and Accountability Commission).

Specific Aims for Follow-up Survey:

The goal of the follow-up survey, to be conducted 4-6 weeks after patients have completed their initial website review and their initial survey, is to explore impacts in terms of use of services, and effects on mental health stigma and brief measures of stress/anxiety, and provide follow-up information on mediating factors such as experience of stress including with the COVID-19 pandemic. The follow-up survey will provide evaluative data on somewhat longer-term impact than the immediate quantitative survey.

Specific Aim 5: To understand the experience of users who reviewed the website of free mental health resources, 4-6 weeks after their initial survey.

Specific Aim 6: To understand any associations of experience of the website with mental health stigma items, and use of services; as well as any continued use of the website resources; and explore changes in risk for depression and anxiety (PHQ2 and GAD2) and context for stresses due to the COVID-19 pandemic.

Linkage to Survey and Google Analytics Data for follow-up survey Survey data will also be linked to respondents' initial survey and google analytics data, to understand the context of website use and user characteristics for the sample.

ELIGIBILITY:
Inclusion Criteria: Participants must be:

* 18 years or older by self-report
* able to access the internet on their own
* able to complete a written survey in English or Spanish.
* They must be invited by a partnering agency within the limit allowed to that agency (30-40 participants).

Exclusion Criteria:

* Age under 18 by self-report
* inability to read and understand either English or Spanish
* not having access online (not a specific survey question).
* Not able to complete survey in English or Spanish;
* Referring stakeholder group has already had 30-40 participants enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (>=18) that partner with agencies participating across California in the evaluation of the Together for Wellness website, and voluntarily agree to participate. This will include community members, community leaders, case managers and crisis counselors, and clients of agencies.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2023-01-07 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-2 item (PHQ-2) | change from baseline to 4-6 weeks follow-up
  Screener for depressive disorder
Generalized Anxiety Disorder-2 items (GAD-2) | change from baseline to 4-6 weeks follow-up
  Screener for generalized anxiety disorder

SECONDARY OUTCOMES:
Stigma toward mental health | change from baseline to 4-6 weeks follow-up
  2-item measure (5 agree to disagree categories plus don't know)
Behavioral Health Services Use | Change from baseline to 4-6 weeks follow-up
  ER use, general medical use, mental health provider use, substance use provider use, hospitalization for behavioral health, residential treatment, hotline use for behavioral health (any, visits/nights/calls if any, for ER use and general medical also visits for behavioral health); -- overall: any use, mean visits and for behavioral health visits
COVID-related Stressors | Change from baseline to 4-6 weeks follow-up
  Pandemic stress index (adapted):
  Overall impact (5 categories plus not answer); experience of stressors (18 plus other)
Race/ethnicity discrimination | Change from baseline to 4-6 weeks follow-up
  race/ethnicity discrimination measure (6 items on 4-point agree scale)
vaccination status and acceptability | Change from baseline to 4-6 weeks follow-up
  vaccination status (yes/no) and acceptability (5 category agree, plus don't know)
perceived value of website | Change from baseline to 4-6 week follow-up
  Baseline: Satisfaction, ease of use, relevance (4-items, 5 agree categories plus don't know); mean
  Follow-up: any use (yes/no); frequency of use/download (4 categories); use and value of 6 resources areas (any use; 4 categories of value if used); recommended site to others (yes/no; how many times open ended; which categories of 6- any use (0/1) frequency (count) and by category

CONTACTS AND LOCATIONS:
Overall Officials: MarySue Heilemann, PhD, Study Director — UCLA School of Nursing
Locations (1):
- UCLA Jane and Terry Semel Institute for Neuroscience and Human Behavior, Center for Health Services and Society, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
The data will be deidentified and linked by code number; we will be deciding whether deidentified data will be available to other investigators from this pilot study.

REFERENCES:
- [Result] Wells K, Thames AD, Young AS, Zhang L, Heilemann MV, Romero DF, Oliva A, Jones F, Tang L, Brymer M, Elliott T, Arevian A; Together for Wellness/Juntos Collaborators and Writing Group. Engagement, Use, and Impact of Digital Mental Health Resources for Diverse Populations in COVID-19: Community-Partnered Evaluation. JMIR Form Res. 2022 Dec 7;6(12):e42031. doi: 10.2196/42031. PMID 36346902